CLINICAL TRIAL: NCT00754247
Title: A Prospective, Randomized, Investigator-blinded, Placebo-controlled, Comparative Study Evaluating the Tolerability and Efficacy of Two Topical Therapies for the Treatment of Keloids and Hypertrophic Scars
Brief Title: A Randomized Comparative Study Evaluating the Tolerability and Efficacy of Two Topical Therapies for the Treatment of Keloids and Hypertrophic Scars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20060131
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Keloid; Hypertrophic Scar; Cicatrix, Hypertrophic
Keywords: Keloid; Hypertrophic scar; Hydrocortisone, silicone, vitamin E lotion; HSE; Onion extract gel; OE; Cetearyl alcohol lotion; CEA
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic | interventions — Hydrocortisone; Silicones; Ethanol; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen A (Experimental): 0.5% hydrocortisone, silicone, vitamin E lotion
  Interventions: Drug: 0.5% hydrocortisone, silicone, vitamin E lotion
- Regimen B (Experimental): Onion extract gel
  Interventions: Drug: Onion extract gel
- Regimen C (Placebo Comparator): Cetearyl alcohol lotion
  Interventions: Drug: Cetearyl alcohol lotion

INTERVENTIONS:
Drug: 0.5% hydrocortisone, silicone, vitamin E lotion — 0.5% hydrocortisone, silicone, vitamin E lotion will be applied topically to cover the selected scar twice daily for 16 weeks. The lesion will be cleansed with soap and water and dried thoroughly. The medication will be applied with a brush and allow it to dry for one minute before contact with clothing.
  Other Names: Scarguard
  Arms: Regimen A
Drug: Onion extract gel — Onion extract gel is applied and massaged into the selected scar 3 to 4 times daily according to product instructions for 16 weeks.
  Other Names: Mederma
  Arms: Regimen B
Drug: Cetearyl alcohol lotion — Placebo is cetearyl alcohol lotion with no steroids, silicone, vitamin E, or onion extract and will be applied 2 times a day to the lesion.
  Other Names: Cetaphil lotion
  Arms: Regimen C

SUMMARY:
Keloids are thought to result from derailments in the typical wound healing process following cutaneous injury. Current treatment options for keloids include intralesional corticosteroids, silicone gel sheeting, compression, surgery and adjuvants to surgery, including radiation and cryotherapy.

0.5% hydrocortisone, silicone, vitamin E lotion (HSE) and onion extract gel (OE) are widely used over-the-counter medications for the treatment of keloids and hypertrophic scars. However, their efficacy and safety have not been compared in a blinded, placebo-controlled, prospective fashion. This study is being undertaken to determine the efficacy and safety of HSE versus OE versus placebo (Cetearyl alcohol; CEA) in subjects with hypertrophic scars and keloids.

This is an investigator-blinded study, which means that the doctor evaluating you will not know if you are receiving the study medication or not. Another doctor will be supplying you with the medication and discussing any problems that you may have with the medication.

You will be assigned to one of the three treatment groups: HSE, OE, or CEA. The group will be assigned by chance and you will have two in three chances of receiving treatment with a study medication, HSE or OE. The no treatment group will receive CEA, a bland lotion, containing no active ingredients such as steroids, silicone, vitamin E, or onion extract.

DETAILED DESCRIPTION:
This study will last up to 16 weeks, with a total of 5 visits to the clinic (Baseline visit, Week 4, 8, 12, and 16 ), excluding the Screening Visit.

Screening Visit/Baseline Visit:

Patients will read and be explained the informed consent. Patients who agree to participate will sign the informed consent and a copy will be given to them. Medical history and exclusion/inclusion criteria will be reviewed; if a patient qualifies he/she will be assigned a randomization number for the treatment.

At the baseline visit, medical history and exclusion/inclusion criteria since the screening visit will be reviewed. Patients randomized to the HSE group will receive one tube and apply the first application to the keloid/hypertrophic scar during the baseline visit. Patients randomized to the OE group will be given a tube of OE gel and will apply the first application to the keloid/hypertrophic scar. Patients in the placebo group will be given a bottle of CEA lotion, the placebo medication, and will apply the first application to the keloid/hypertrophic scar. The medications will be given by the unblinded investigator and the blinded investigator will be evaluating the patients. Photographs of the patient's keloid/hypertrophic scar will be taken, and the keloid/hypertrophic scar will be measured/assessed according to Methods of Study Lesion Assessment (below). A urine pregnancy test will be obtained for all women of child-bearing potential.

Week 4, 8, 12, and 16 Visit:

Patients will be asked about side effects since last visit. Photographs of the patient's keloid/hypertrophic scar will be taken and the keloid/hypertrophic scar will be measured/assessed according to Methods of Study Lesion Assessment (below). A urine pregnancy test will be obtained at for all women of child-bearing potential.

Methods of Study Lesion Assessment

A. Volume B. Linear dimensions

Investigator's Assessments w/ Visual Analog Scale (VAS):

C. Cosmetic assessment D. Induration (hardness) [compared to standardized hard discs with numerical ranking of increased induration] E. Erythema (redness) F. Pigmentary alteration

Patient's Assessments w/ VAS:

G. Cosmetic assessment H. Pain I. Tenderness J. Pruritus (itching) K. Patient satisfaction

L. Digital photographs

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Male or female, at least 18 years old in good general health, that have a hypertrophic and keloid scar. The length of the scar should be between 1-4 cm. Individuals who are willing and able to follow the requirements for study participation
2. The investigator believes that the scar could benefit from the study medication.

Exclusion Criteria:

Subjects who meet any of the following criteria should be excluded from the study:

1. Individuals with target scar that is not amenable to the randomized treatment
2. Individuals who are planning pregnancy, or pregnant as determined by urine pregnancy test during the duration of the study, or breast-feeding an infant
3. Individuals with uncontrolled diabetes or autoimmune disorders
4. Individuals who have received scar treatment within one month of the first day of study treatment
5. Individuals who plan to receive scar treatment(s) other than study treatment during the trial
6. Individuals with a known sensitivity to any ingredients in the test products
7. Individuals with any skin conditions or taking any medications that may interfere with the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, M.D., Ph.D, Principal Investigator — University of Miami, Department of Dermatology and Cutaneous Surgery
Locations (1):
- University of Miami Skin Research Group Office, Miami, Florida, United States

REFERENCES:
- [Background] Augusti KT. Therapeutic values of onion (Allium cepa L.) and garlic (Allium sativum L.). Indian J Exp Biol. 1996 Jul;34(7):634-40. PMID 8979497
- [Background] Saulis AS, Mogford JH, Mustoe TA. Effect of Mederma on hypertrophic scarring in the rabbit ear model. Plast Reconstr Surg. 2002 Jul;110(1):177-83; discussion 184-6. doi: 10.1097/00006534-200207000-00029. PMID 12087249
- [Background] Musgrave MA, Umraw N, Fish JS, Gomez M, Cartotto RC. The effect of silicone gel sheets on perfusion of hypertrophic burn scars. J Burn Care Rehabil. 2002 May-Jun;23(3):208-14. doi: 10.1097/00004630-200205000-00010. PMID 12032371
- [Background] Phillips TJ, Gerstein AD, Lordan V. A randomized controlled trial of hydrocolloid dressing in the treatment of hypertrophic scars and keloids. Dermatol Surg. 1996 Sep;22(9):775-8. doi: 10.1111/j.1524-4725.1996.tb00728.x. PMID 8874525
- [Background] Eisen D. A pilot study to evaluate the efficacy of scarguard in the prevention of scars. Internet J Dermatol. 2004;5.
- [Background] Gilman TH. Silicone sheet for treatment and prevention of hypertrophic scar: a new proposal for the mechanism of efficacy. Wound Repair Regen. 2003 May-Jun;11(3):235-6. doi: 10.1046/j.1524-475x.2003.11313.x. No abstract available. PMID 12753606
- [Background] Jackson BA, Shelton AJ. Pilot study evaluating topical onion extract as treatment for postsurgical scars. Dermatol Surg. 1999 Apr;25(4):267-9. doi: 10.1046/j.1524-4725.1999.08240.x. PMID 10417579
- [Background] Chung VQ, Kelley L, Marra D, Jiang SB. Onion extract gel versus petrolatum emollient on new surgical scars: prospective double-blinded study. Dermatol Surg. 2006 Feb;32(2):193-7. doi: 10.1111/j.1524-4725.2006.32045.x. PMID 16442038
- See also: Skin Research Group Website — http://www.skininvestigation.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Detailed enrollment data for participants is not available for week 4, 8, and 12.
  Reason participants did not complete study are not available for reporting.
Groups:
- 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ): 0.5% hydrocortisone, silicone, vitamin E lotion
  0.5% hydrocortisone, silicone, vitamin E lotion: 0.5% hydrocortisone, silicone, vitamin E lotion will be applied topically to cover the selected scar twice daily for 16 weeks. The lesion will be cleansed with soap and water and dried thoroughly. The medication will be applied with a brush and allow it to dry for one minute before contact with clothing.
- Onion Extract Gel (OE): Onion extract gel
  Onion extract gel: Onion extract gel is applied and massaged into the selected scar 3 to 4 times daily according to product instructions for 16 weeks.
- Cetearyl Alcohol Lotion (Placebo): Cetearyl alcohol lotion
  Cetearyl alcohol lotion: Placebo is cetearyl alcohol lotion with no steroids, silicone, vitamin E, or onion extract and will be applied 2 times a day to the lesion.
Period: Overall Study
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Started | 10 | 10 | 10
Completed | 5 | 5 | 5
Not Completed | 5 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are available for the 15 participants that completed the week 16 visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Lesion Volume
Description: Blinded investigator assessed the scar volume by using an alginate impression.
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent Change | 40 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 42 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 32 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

2. Secondary Outcome: Change in Lesion Length
Description: Blinded investigator assessed the scar length. Measured with ruler, from scar tip to tip.
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent change | 12 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 13 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 3 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

3. Secondary Outcome: Change in Lesion Width
Description: Blinded investigator assessed the scar width. Measured with a ruler at the visually largest width.
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent change | 0 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 16 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 5 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

4. Secondary Outcome: Change in Lesion Induration
Description: Blinded investigator assessed the scar induration. Measured with a ruler at deepest point.
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent change | 68 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 50 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 2 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

5. Secondary Outcome: Change in Lesion Erythema
Description: Blinded investigator assessed the scar erythema. Measured with a visual analog scale (VAS), ranging from 0-100 (0=best and 100=worst).
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent change | 72 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 8 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 1 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

6. Secondary Outcome: Change in Lesion Pigmentary Alteration
Description: Blinded investigator assessed the scar pigmentation alteration using a visual analog scale (VAS), ranging from 0-100 (0=best and 100=worst).
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent change | 61 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 30 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 0 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

7. Secondary Outcome: Change in Lesion Cosmetic Appearance
Description: Blinded investigator assessed the scar cosmetic appearance using a visual analog scale (VAS), ranging from 0-100 (0=best and 100=worst).
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent change | 68 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 25 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 15 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

8. Secondary Outcome: Change in Lesion Cosmetic Appearance
Description: Subjects assessed the scar cosmetic appearance with a visual analog scale (VAS), ranging from 0-100 (0=best and 100=worst).
Time Frame: Assessed at Baseline visit (week 0) and week 16
Population: Data only available for participants that completed week 16 visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
Number analyzed (Participants) | 5 | 5 | 5
Percent change | 48 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 20 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 58 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

ADVERSE EVENTS:
Time Frame: Week 16
Arm/Group | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) | Onion Extract Gel (OE) | Cetearyl Alcohol Lotion (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5% Hydrocortisone, Silicone, Vitamin E Lotion (HSE ) (N=10) | Onion Extract Gel (OE) (N=10) | Cetearyl Alcohol Lotion (Placebo) (N=10)
Acneiform-like eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes